CLINICAL TRIAL: NCT00937755
Title: The Study of Atypical Antipsychotics-induced Metabolic Disturbances
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Other Study IDs: F941101
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Schizophrenia; Antipsychotics
Keywords: schizophrenia; antipsychotics; glucose homeostasis; metabolic disturbance
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- olanzapine: olanzapine 10-20 mg/day
- quetiapine: quetiapine 300-600 mg/day
- risperidone: risperidone monotherapy, 2-4 mg/day

SUMMARY:
Schizophrenia is one of the most severe mental illnesses. The antipsychotic drugs, introduced in early 1950s, have revolutionized the treatment of schizophrenia. About 2 to 4 times as many patients relapse when treated with a placebo as do those treated with antipsychotic drugs. For these medications to be maximally beneficial, they must have an acceptable side effect profile and be taken as prescribed. One untoward effect of many antipsychotic drugs is weight gain. The extent of weight gain apparently varies by drug, which may be because of drugs'differing degrees of action on serotonergic, dopaminergic, histaminergic, and other neurotransmitter systems. Obesity is a threat to health and longevity. Weight gain may also cause patients taking antipsychotic medication to discontinue their medication, which may predispose them to relapse.

The pattern of weight gain and metabolic disturbance may vary between the different antipsychotic agents. The underlying mechanism and treatment of these adverse metabolic effects remain unclear. This study will recruit 60 schizophrenic patients during. The patients received monotherapy with atypical antipsychotics (olanzapine, quetiapine, or risperidone). The assessment of metabolic profile will be monitored at baseline, week 2, week 4, and week 8. The measurements include anthropometrical parameters, body composition, glucose level, insulin level, lipid profile, and leptin level. Intra-venous glucose tolerance test will be used to assess the insulin secretion and insulin sensitivity.

This proposal broadly aims to discover the underlying mechanism of antipsychotics induced metabolic disturbance and develop efficient treatment to correct it.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of schizophrenia
* age 18-60 years

Exclusion Criteria:

* received any SGAs prior to this study
* medical conditions that may confound glucoregulatory assessment
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: psychiatric outpatient clinic and inpatient units
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
glucose homeostasis | 8 weeks

SECONDARY OUTCOMES:
lipid homeostasis | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University-Municipal Wan-Fang Hospital, Taipei, Taiwan